CLINICAL TRIAL: NCT04669730
Title: Baduanjin Exercise on Lung Operative
Brief Title: Baduanjin Exercise on Meridian Energy, Lung Function and Heart Rate Variability in Patients Undergoing Lung Operative.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Chun Hou Huang, Assistance Professor, Tzu Chi University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: TCU-CHHuang-BaduanjinLungCa
Record Dates: First submitted 2020-11-29; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Lung Cancer Non Small Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Walking

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm A: usual care (Placebo Comparator): Routine usual care
  Interventions: Other: usual care
- Arm B: walk (Active Comparator): Walk 30mins per day, 5 days per week.
  Interventions: Behavioral: Walk
- Arm C: Baduanjin (Active Comparator): Baduanjin 12 mins per day, 5 days per week.
  Interventions: Behavioral: Baduanjin
- Arm D: Baduanjin plus walk (Experimental): Walk 30mins then Baduanjin 12 mins per day, 5 days per week.
  Interventions: Behavioral: Baduanjin plus walk

INTERVENTIONS:
Other: usual care — Routine care
  Arms: Arm A: usual care
Behavioral: Walk — Walk 30mins
  Arms: Arm B: walk
Behavioral: Baduanjin — Baduanjin exercise is moderate in intensity and short in duration (a set of Baduanjin takes about 12 minutes). Baduanjin consists of the sitting and standing practicing form. The sitting Baduanjin exercise conforms to the aspects of low-intensity and long-term aerobic activity, which is suitable for the rehabilitation training of patients who are in stable condition during hospitalization. The standing Baduanjin is more suitable for patients with sequential rehabilitation after discharge and can be adjusted based on the patient's condition
  Arms: Arm C: Baduanjin
Behavioral: Baduanjin plus walk — Walk 30mins then Baduanjin 12mins per day, 5 times per week.
  Arms: Arm D: Baduanjin plus walk

SUMMARY:
Lung cancer (LC) is the leading cause of cancer-related death and is the most frequent cancer in both sexes.Respectable lung tumor with abnormal lung function, usually because of tobacco use, have chronic obstructive pulmonary disease (COPD), coronary artery disease, and/or old age as underlying comorbidities. Until recent, most exercise prescribed using aerobic exercise programs. Baduanjin is a type of movement-based mind-body intervention. It is a form of traditional practice designed to promote physical and psychological health, manage symptoms, and relieve stress during illness. The impacts of a Baduanjin exercise-based cardiopulmonary rehabilitation program for patients recovering from respectable lung tumor on Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan), lung function and heart rate variability has yet to be assessed. This trial evaluates whether the Baduanjin exercise would provide effective lung function, meridian energy and HRV in patients following lung operative.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary NSCLC based on preoperative pathologic examination
* Had no surgical contraindication to and were willing to undergo video-assisted thoracic surgery or traditional thoracotomy (open) lobectomy
* Agreed to receive exercise performed.

Exclusion Criteria:

* SpO2 <90% during the 6-min walking test
* With an absence of NSCLC, as confirmed by postoperative pathologic examination or with sub-lobar resection or pneumonectomy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-05-27 (Estimated); Study Completion 2022-11-27 (Estimated)

PRIMARY OUTCOMES:
The 24 points skin electric conductance over bilateral wrist and foot in patients undergoing lung operative, after admission baseline evaluation before lung operative as assessed using M.E.A.D (Meridian Energy Analysis Device)：Baseline | Baseline
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current. Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing lung operative as assessed using M.E.A.D (Meridian Energy Analysis Device)：2 weeks | 2 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current. Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing lung operative as assessed using M.E.A.D (Meridian Energy Analysis Device)：4 weeks | 4 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current. Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing lung operative as assessed using M.E.A.D (Meridian Energy Analysis Device)：12 weeks | 12 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current. Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.
The change of 24 points skin electric conductance over bilateral wrist and foot in patients undergoing lung operative as assessed using M.E.A.D (Meridian Energy Analysis Device)：16 weeks | 16 weeks
  The electrical conductance of the acupuncture points of human subject can be measured by a computerized testing instrument with a very low electrical current. Ryodoraku theory has been shown to be a supplementary diagnostic method for selective diseases and a useful parameter for evaluating therapeutic effects of acupuncture. The electrical conductance of an acupoint was measured using a Meridian Energy Analysis Device (MEAD100, Med- Pex Enterprises, Taichung, Taiwan) operating at DC 12V and 0 to 200A. The method and procedure of the MEAD is based on the Ryodoraku theory and is similar to equipment used in previous studies.

CONTACTS AND LOCATIONS:
Overall Officials: Chun Hou Huang, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Taiwan